CLINICAL TRIAL: NCT02300129
Title: Effect of CD07805/47 Gel in Subjects Presenting With Flushing Related to Erythematotelangiectatic or Papulopustular Rosacea
Brief Title: Effect of CD07805/47 Gel in Rosacea Flushing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.40225E
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-08

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo (Experimental): Period 1:
  Application of 1g of CD07805/47 0.5% Gel on full face on Day 1 (cross-over design) and 500mg on a half-face (split-face design) on Day 3.
  Application of 500mg of Placebo Gel on a half-face (split-face design) on Day 3 and 1g on full face on Day 5 (cross-over design)
  Period 2 (cross-over design):
  Application of 1g of CD07805/47 0.5% Gel on full face once daily 7 days per week for 2 weeks then 1g of Placebo Gel on full face once daily 7 days per week for 2 weeks
  Interventions: Drug: CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo
- Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo (Experimental): Period 1:
  Application of 1g of Placebo Gel on full face on Day 1 (cross-over design) and 500mg on a half-face (split-face design) on Day 3.
  Application of 500mg of CD07805/47 0.5% Gel on a half-face (split-face design) on Day 3 and 1g on full face on Day 5 (cross-over design).
  Period 2 (cross-over design):
  Application of 1g of CD07805/47 0.5% Gel on full face once daily 7 days per week for 2 weeks then 1g of Placebo Gel on full face once daily 7 days per week for 2 weeks.
  Interventions: Drug: Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo
- CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47 (Experimental): Period 1:
  Application of 1g of CD07805/47 0.5% Gel on full face on Day 1 (cross-over design) and 500mg on a half-face (split-face design) on Day 3.
  Application of 500mg of Placebo Gel on a half-face (split-face design) on Day 3 and 1g on full face on Day 5 (cross-over design).
  Period 2 (cross-over design):
  Application of 1g of Placebo Gel on full face once daily 7 days per week for 2 weeks then 1g of CD07805/47 0.5% Gel on full face once daily 7 days per week for 2 weeks.
  Interventions: Drug: CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47
- Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47 (Experimental): Period 1:
  Application of 1g of Placebo Gel on full face on Day 1 (cross-over design) and 500mg on a half-face (split-face design) on Day 3.
  Application of 500mg of CD07805/47 0.5% Gel on a half-face (split-face design) on Day 3 and 1g on full face on Day 5 (cross-over design).
  Period 2 (cross-over design):
  Application of 1g of Placebo Gel on full face once daily 7 days per week for 2 weeks then 1g of CD07805/47 0.5% Gel on full face once daily 7 days per week for 2 weeks.
  Interventions: Drug: Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47

INTERVENTIONS:
Drug: CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo — Period 1:
  1g of CD07805/47 0.5% Gel on full face on Day 1 and 500mg on a half-face on Day 3.
  500mg of Placebo Gel on a half-face on Day 3 and 1g on full face on Day 5.
  Period 2:
  1g of CD07805/47 0.5% Gel on full face once daily 7 days per week for 2 weeks.
  1g of Placebo Gel on full face once daily 7 days per week the 2 following weeks.
  Arms: CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo
Drug: Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo — Period 1:
  1g of Placebo Gel on full face on Day 1 and 500mg on a half-face on Day 3.
  500mg of CD07805/47 0.5% Gel on a half-face on Day 3 and 1g on full face on Day 5.
  Period 2:
  1g of CD07805/47 0.5% Gel on full face once daily 7 days per week for 2 weeks.
  1g of Placebo Gel on full face once daily 7 days per week the 2 following weeks.
  Arms: Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo
Drug: CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47 — Period 1:
  1g of CD07805/47 0.5% Gel on full face on Day 1 and 500mg on a half-face on Day 3.
  500mg of Placebo Gel on a half-face on Day 3 and 1g on full face on Day 5.
  Period 2:
  1g of Placebo on full face once daily 7 days per week for 2 weeks.
  1g of CD07805/47 0.5% Gel on full face once daily 7 days per week the 2 following weeks.
  Arms: CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47
Drug: Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47 — Period 1:
  1g of Placebo Gel on full face on Day 1 and 500mg on a half-face on Day 3.
  500mg of CD07805/47 0.5% Gel on a half-face on Day 3 and 1g on full face on Day 5.
  Period 2:
  1g of Placebo on full face once daily 7 days per week for 2 weeks.
  1g of CD07805/47 0.5% Gel on full face once daily 7 days per week the 2 following weeks.
  Arms: Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47

SUMMARY:
Phase 2a study to assess the efficacy and safety of CD07805/47 0.5% gel in the prevention of the flush of rosacea.

DETAILED DESCRIPTION:
The objectives of this study in rosacea patients (type I&II) are:

* to demonstrate objectively that CD07805/47 0.5% gel is able to prevent a flush induced by a specific trigger (hot water) in controlled condition;
* to demonstrate that CD07805/47 0.5% gel is able to prevent a flush whatever the trigger in everyday life condition;
* to investigate if reduction in redness is associated with a decrease in skin sensations such as heat, stinging/burning, skin tension and sweating;
* to demonstrate that such efficacy on transient redness and sensations takes place in both populations (rosacea type I and rosacea type II).

This is a single-centre, randomized, Investigator masked, placebo controlled study comprising the following periods:

A screening period of maximum 4 weeks

A one-week treatment phase (Period 1) with 3 sessions using the flush model, every other day.

This Period 1 includes a cross-over design (first and third sessions) and a split face design (second session). During this period, thirty six (36) subjects will receive on site the study drugs as follows (the order of each session being randomized):

* CD07805/47 placebo gel on both sides of the face,
* one side of the face treated with CD07805/47 0.5% gel, the other side treated with the CD07805/47 placebo gel (the allocation of treatment on each half-face will be determined according to a randomization list),
* CD07805/47 0.5% gel on both sides of the face;

A 2-days wash-out period (between Period 1 and Period 2) with no treatment on either side of the face

A 4-week treatment phase (Period 2) corresponding to a cross-over design during which the subjects will apply themselves the study drugs at home on the whole face, once daily 7 days per week.

The subjects will be divided in 2 groups of eighteen (18) subjects and will receive either the CD07805/47 0.5% gel the first 2 weeks and then the CD07805/47 placebo gel or the CD07805/47 placebo gel the first 2 weeks and then the CD07805/47 0.5% gel, according to randomization.

All the subjects taking part into the study will not be randomized separately in the two periods but to the full sequence at the beginning of the clinical trial (same randomization number during all the study), explaining the arms/groups detailed in the section "Arms and Interventions".

Only primary efficacy endpoint: total number of flushes for each 2-week period will be detailed in the outcome measures section.

The other endpoints are secondary or exploratory.

The purpose of Period 1 is to assess whether simpler and shorter designs based on flush induced by a trigger could be as efficient to detect prevention of flush than the more classical and longer design of Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or female, who is at least 18 years of age or older at Screening visit.
2. The subject has a clinical diagnosis of mild to moderate erythemato-telangiectatic rosacea or mild to moderate papulo-pustular rosacea according to the National Rosacea Society grading (Wilkin et al., 2004)
3. The subject had at least five flushing episodes during the last week before Screening and Baseline visits

Exclusion Criteria:

1. The subject has particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin), or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus or actinic telangiectasia;
2. The subject has current treatment with monoamine oxidase inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, or alpha-agonists;
3. The subject has less than 3 months stable dose treatment with tricyclic anti-depressants, cardiac glycosides, beta blockers or other antihypertensive agents;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Galderma Investigational site, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo: Period 1:
  Application of 1g of CD07805/47 0.5% Gel on full face on Day 1 (cross-over design) and 500mg on a half-face (split-face design) on Day 3.
  Application of 500mg of Placebo Gel on a half-face (split-face design) on Day 3 and 1g on full face on Day 5 (cross-over design).
  Period 2 (cross-over design):
  Application of 1g of CD07805/47 0.5% Gel on full face once daily 7 days per week for 2 weeks then 1g of Placebo Gel on full face once daily 7 days per week for 2 weeks.
Period: Period 1 Session 1 (Day 1)
Arm/Group | CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo | Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo | CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47 | Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47
Started | 11 | 5 | 7 | 11
Completed | 11 | 5 | 7 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Period 1 Session 2 (Day 3)
Arm/Group | CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo | Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo | CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47 | Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47
Started | 11 | 5 (Withdrawal consent of 1 subject between Day 1 and Day 3) | 7 | 11
Completed | 11 | 4 | 7 | 11
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Period 1 Session 3 (Day 5)
Arm/Group | CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo | Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo | CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47 | Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47
Started | 11 | 4 | 7 | 11
Completed | 11 | 4 | 7 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 Treatment 1 (2 Weeks)
Arm/Group | CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo | Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo | CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47 | Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47
Started | 11 | 4 | 7 | 11 (Withdrawal consent of 1 subject between the Period 1 and Period 2)
Completed | 10 | 4 | 7 | 10
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Period 2 Treatment 2 (2 Weeks)
Arm/Group | CD07805/47, CD07805/47+Placebo, Placebo, CD07805/47, Placebo | Placebo, CD07805/47+Placebo, CD07805/47, CD07805/47, Placebo | CD07805/47, CD07805/47+Placebo, Placebo, Placebo, CD07805/47 | Placebo, CD07805/47+Placebo, CD07805/47, Placebo, CD07805/47
Started | 10 | 4 | 7 | 10
Completed | 10 | 4 | 7 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat population
Groups:
- All Study Participants (Intent To Treat Population): One subject was excluded from Intent to Treat (ITT) population because he didn't perform any efficacy assessment during the study so N=33 instead of 34 subjects
Arm/Group | All Study Participants (Intent To Treat Population)
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 2
Region of Enrollment [Number; unit: participants]
  Germany | 33

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Flushes for Each 2-week Period
Time Frame: Day 22 and Day 36/Early termination
Population: Per protocol population of Period 2, N= 31
Measure: Mean (Standard Deviation); unit: Flushes count
Groups:
- Period 2 CD07805/47 0.5% Gel Cross-over: CD07805/47 0.5% gel (Brimonidine tartrate)
- Period 2 Placebo Gel Cross-over: CD07805/47 placebo gel
Arm/Group | Period 2 CD07805/47 0.5% Gel Cross-over | Period 2 Placebo Gel Cross-over
Number analyzed (Participants) | 31 | 31
Flushes count | 15.3 (12.1) | 16.3 (14.0)
Statistical Analysis 1: Comparison: Period 2 CD07805/47 0.5% Gel Cross-over vs Period 2 Placebo Gel Cross-over; Test type: Superiority or Other; p = 0.7420, ANOVA — P value associated to treatment effect in the model. Study design with a power of 80% and a type I error at 5% (two-sided); Analysis of variance including sequence, subject (sequence), period and treatment as factors in the model

ADVERSE EVENTS:
Groups:
- Period 1 Placebo Gel Cross Over: Period 1 Placebo gel cross over (application on full face) Overall safety population, N=34
- Period 1 CD07805/47 0.5% Gel Split Face: Period 1 CD07805/47 0.5% gel split face (application on one side of face) Overall safety population, N=33
- Period 1 Placebo Gel Split Face: Period 1 Placebo gel split face (application on one side of face) Overall safety population, N=33
- Period 1 CD07805/47 0.5% Gel Cross-over: Period 1 CD07805/47 0.5% cross over (application on full face) Overall safety population, N=33
- Period 2 CD07805/47 0.5% Gel Cross Over: Period 2 CD07805/47 0.5% gel (application on full face) Overall safety population, N=32
- Period 2 Placebo Gel Cross Over: Period 2 Placebo gel cross over (application on full face) Overall safety population, N=31
Arm/Group | Period 1 Placebo Gel Cross Over | Period 1 CD07805/47 0.5% Gel Split Face | Period 1 Placebo Gel Split Face | Period 1 CD07805/47 0.5% Gel Cross-over | Period 2 CD07805/47 0.5% Gel Cross Over | Period 2 Placebo Gel Cross Over
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/33 | 0/33 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 2/33 | 1/33 | 4/32 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Placebo Gel Cross Over (N=34) | Period 1 CD07805/47 0.5% Gel Split Face (N=33) | Period 1 Placebo Gel Split Face (N=33) | Period 1 CD07805/47 0.5% Gel Cross-over (N=33) | Period 2 CD07805/47 0.5% Gel Cross Over (N=32) | Period 2 Placebo Gel Cross Over (N=31)
Erythema and skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Cutaneous AE related to CD07805/47 0.5% gel
Erythema, papules and pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) — Cutaneous AE related to CD07805/47 placebo gel
Erythema, papules and pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) — AE of Special Interest related to CD07805/47 0.5% gel leading to subject discontinuation
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Cutaneous AE not related to CD07805/47 0.5 gel
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Cutaneous AE not related to CD07805/47 0.5 gel
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) — Cutaneous AE not related to CD07805/47 0.5 gel
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non cutaneous AE
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non cutaneous AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other